CLINICAL TRIAL: NCT06117293
Title: Safety and Efficacy Evaluation of the Mosaic Ultra Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CynosureLutronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMI22001
Record Dates: First submitted 2023-10-23; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Skin Texture Disorder; Photoaging; Wrinkle; Scar; Stretch Mark; Acne Vulgaris; Hair Loss
MeSH Terms: conditions — Cicatrix; Striae Distensae; Acne Vulgaris; Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Subjects will be treated up to 5 times with a 30- and 90-day post final-treatment follow-up. Subjects may be asked to participate in an elective biopsy collected from normal skin simultaneously.
  Interventions: Device: Mosaic

INTERVENTIONS:
Device: Mosaic — 1550 Fractional Laser System

SUMMARY:
Evaluate the Safety and Efficacy of the Mosaic Ultra 1550nm system for the treatment of skin tone and texture, facial rejuvenation, photoaging, wrinkles, scars, stretch marks, acne vulgaris and hair loss.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, Male or Female
* Age 18 - 60 years old
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated.
* Participants who are willing and able to comply with all study participation requirements including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* OPTIONAL - Participants who are willing to undergo biopsies.

Exclusion Criteria:

* Previous surgical or cosmetic procedure to the target area in the last 6 to 12 months that could interfere with the treatment procedure
* A study participant must not be pregnant or have been pregnant in the last 3 months
* A recent history of smoking (6 months)
* Presence of an active skin disease or condition that may affect wound healing (ie. diabetes myelitis; connective tissue disease; radiation therapy; or chemotherapy)
* Seizure disorder caused by bright light
* A history of thrombophlebitis
* A history of acute infections
* A history of heart failure
* Cancer, malignant disease, skin pathology, condition, or allergic reactions that could interfere with evaluation or with the use of typical ancillary medical treatments or care used before, during, or after treatments
* Received or is anticipated to receive antiplatelets, anticoagulants, thrombolytics, vitamin E, or anti-inflammatories within 2 weeks prior to treatment
* Intolerance or allergy to medications that could be prescribed before or after the procedure (eg, antibiotics, anesthesia)
* A history of keloids
* A history or evidence of poor wound healing
* A history of coagulative disorder or current use of anticoagulant drugs within 2 weeks of study participation
* Use of steroids within 2 weeks of study treatments
* Patients with implanted pacemaker or defibrillator, or metal pins, or prosthetic joints within 4 cm of treatment area
* History of psychoneurosis and/or a history of alcohol or drug abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Photographic Assessment | 90-day Follow-Up
  Evaluation of Randomized Before Treatment and 3-Month Follow-Up Images by Blinded Evaluators

SECONDARY OUTCOMES:
Safety Assessment | up to 90 days post final treatment
  Evaluation of Adverse Events
Subject Satisfaction | 30-day and 90-day Follow-Up
  Scoring of Satisfaction from Extremely Satisfied to Extremely Dissatisfied
Physician Satisfaction | 30-day and 90-day Follow-Up
  Scoring of Satisfaction from Extremely Satisfied to Extremely Dissatisfied
Subject Clinical Global Aesthetic Improvement Scale | 30-day and 90-day Follow-Up
  Scoring on the Clinical Global Aesthetic Improvement Scale is completed by having the subject select one option from the scale corresponding to their perspective of the improvement seen in their treated conditions.
  Response options are 1 - Very Much Improved, 2 - Much Improved, 3 - Improved, 4 - No Change, and 5 - Worsened. A response of 1 - Very Much Improved is the best outcome while a score of 5 - Worsened is the worse outcome.
Physician Clinical Global Aesthetic Improvement Scale | 30-day and 90-day Follow-Up
  Scoring on the Clinical Global Aesthetic Improvement Scale is completed by having the physician select one option from the scale corresponding to their perspective of the improvement seen in their treated conditions of the subject.
  Response options are 1 - Very Much Improved, 2 - Much Improved, 3 - Improved, 4 - No Change, and 5 - Worsened. A response of 1 - Very Much Improved is the best outcome while a score of 5 - Worsened is the worse outcome.
Coagulation Zone Measurements | Baseline, Immediate Post Treatment, 4 Days Post, 14 Days Post, 21 Days Post
  Biopsies taken from healthy tissue prior to treatment up to 21 days post treatment to evaluate histological effect of the device. Tissue samples will be evaluated and the depth and width of the coagulation zones due to the laser (measures in micrometers)
Epidermal Inflammatory Response | Baseline, Immediate Post Treatment, 4 Days Post, 14 Days Post, 21 Days Post
  Biopsies taken from healthy tissue prior to treatment up to 21 days post treatment to evaluate histological effect of the device. Tissue samples will be reviewed for markers of inflammation and coagulation in the epidermis. General comments and observations of the tissue will be completed by a pathologist.
Dermal Inflammatory Response | Baseline, Immediate Post Treatment, 4 Days Post, 14 Days Post, 21 Days Post
  Biopsies taken from healthy tissue prior to treatment up to 21 days post treatment to evaluate histological effect of the device. Tissue samples will be reviewed for markers of inflammation and coagulation in the dermis. General comments and observations of the tissue will be completed by a pathologist.
Tissue Reepithelization | Baseline, Immediate Post Treatment, 4 Days Post, 14 Days Post, 21 Days Post
  Biopsies taken from healthy tissue prior to treatment up to 21 days post treatment to evaluate histological effect of the device. Tissue samples will be evaluated to determine the timepoint in which there is a reepithelization of the treated tissue. Timepoint of reepithelization will be determined by a pathologist reviewing the imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Ibrahimi, Principal Investigator — Lutronic Medical Director
Locations (3):
- United States (3):
  - Advanced Dermatology, Lincolnshire, Illinois
  - Lutronic, Billerica, Massachusetts
  - Dermatology & Skin Health, Peabody, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Plan will not be shared

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT06117293/Prot_SAP_000.pdf